CLINICAL TRIAL: NCT03068728
Title: Analysis of Hemostatic Agents Compared to Physiologic Hemostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Principal Investigator, Jastin Antisdel, MD, Assistant Professor, St. Louis University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24331
Record Dates: First submitted 2017-02-20; First posted 2017-03-03 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Rhino Sinusitis
Keywords: bilateral chronic rhino sinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Intervention Model Description: After sinus surgery, the surgeon will randomize the patient to one of six hemostatic agents and place that product in one sinus cavity, while leaving the other sinus cavity without packing. The treatment group will be compared to control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Study Participants (Other): Participants received hemostatic packing agent in one nasal cavity and no packing in the other.
  Participants were randomized to one of three hemostatic packing agents (Arista, Nexfoam, Nasopore) through sealed envelope, chosen by surgeon prior to placement, with packing agent allocation and sidedness.
  Interventions: Device: Arista; Device: Nexfoam; Device: Nasopore

INTERVENTIONS:
Device: Arista
Device: Nexfoam
Device: Nasopore

SUMMARY:
This study is a prospective comparison between absorbable hemostatic agents as a group and the body's natural hemostatic ability without aid of therapy in patients undergoing bilateral sinus surgery with or without septoplasty.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of absorbable hemostatic agents in comparison with physiologic hemostasis after endoscopic sinus surgery. The investigators aim to determine the relative efficacy of hemostatic agents to halt epistaxis and compare this with the degree of epistaxis observed without therapy and evaluate objective healing parameters.

ELIGIBILITY:
Inclusion Criteria:

-≥18 to <75 years of age with bilateral chronic or recurrent rhino sinusitis recalcitrant to medical therapy that requires endoscopic sinus surgery

-sinuses should have a similar degree of disease involvement bilaterally.

Exclusion Criteria:

* massive sinonasal polyposis,
* history of underlying immunologic diseases, AIDS, cystic fibrosis, immunoglobulin deficiency, immotile cilia syndrome, and neutropenia,
* known hypersensitivity to the aforementioned agents,
* women who are pregnant or breastfeeding,
* anyone with a known allergy to any of the treatments (potato starch, iodine, shellfish)
* anyone with a known coagulopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-05-13 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with superior healing qualities after use of hemostatic agents compared to physiologic hemostasis after endoscopic sinus surgery. | 6 weeks post-operative
  Participants will be monitored for 6 weeks. Means and standard deviations will be obtained for data collected from patient surveys rating subjective symptoms such as nasal obstruction, bleeding, pain, and nasal discharge on a scale ranging from 1-10 and investigator surveys evaluating the qualities of the patient's recovery (synechiae formation, granulation, edema, infection, and time spent debriding the sinuses) in response to intervention and compare this with the degree of epistaxis observed without therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jastin L Antisdel, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT03068728/Prot_SAP_ICF_000.pdf